CLINICAL TRIAL: NCT01614899
Title: Randomized, Double-blind, Parallel- Group, Placebo-controlled, Confirmatory Study of SM-13496 (Lurasidone HCl) in Patients With Schizophrenia <Phase 3>
Brief Title: A Phase III Study of SM-13496 (Lurasidone HCl) in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1001056; JapicCTI-121859 (Registry Identifier: JAPIC Clinical Traials Information)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SM-13496 40mg (Experimental)
  Interventions: Drug: SM-13496 40mg
- SM-13496 80mg (Experimental)
  Interventions: Drug: SM-13496 80mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SM-13496 40mg — once daily orally
  Arms: SM-13496 40mg
Drug: SM-13496 80mg — once daily orally
  Arms: SM-13496 80mg
Drug: Placebo — once daily orally
  Arms: Placebo

SUMMARY:
The study evaluates the efficacy and safety of SM-13496 compared with placebo in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient meets DSM-IV-TR criteria for schizophrenia.
* Patient is aged 18 through 74 years at informed consent.
* Patient understands the objectives, procedures, and possible benefits and risks of the study and who provide written voluntarily consent to participate in the study

Exclusion Criteria:

* Patient has a history of neuroleptic malignant syndrome, water intoxication, or paralytic ileus.
* Patient has Parkinson's disease.
* Patient has a history or complication of malignancy.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2012-07-02; Primary Completion 2014-11-17 (Actual); Study Completion 2014-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Drug development Division, Study Director — Sumitomo Pharma Co., Ltd.
Locations (4):
- 69 Sites, Tokyo, Etc, Japan
- 10 Sites, Kuala Lumpur, Etc, Malaysia
- 22 Sites, Seoul, Etc, South Korea
- 14 Sites, Taipei, Etc, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- SM-13496 (Lurasidone HCl) 40mg: SM-13496 40 mg was administered orally once daily.
- SM-13496 (Lurasidone HCl) 80mg: SM-13496 80 mg was administered orally once daily.
- Placebo: Placebo was administered orally once daily.
Period: Overall Study
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Started | 150 | 155 | 152
Completed | 106 | 116 | 110
Not Completed | 44 | 39 | 42

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo | Total
Number analyzed (Participants) | 145 | 152 | 142 | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (13.1) | 43.6 (13.9) | 42.9 (13.5) | 42.9 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 73 | 58 | 196
  Male | 80 | 79 | 84 | 243
Region of Enrollment [Number; unit: participants]
  Japan | 62 | 66 | 60 | 188
  Taiwan | 19 | 21 | 19 | 59
  Korea, Republic of | 43 | 42 | 43 | 128
  Malaysia | 21 | 23 | 20 | 64

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Positive and Negative Syndrome Scale (PANSS) Total Score at Week 6
Description: The PANSS is an interview-based measure of the severity of psychopathology in adults with psychotic disorders. The measure is comprised of 30 items and three subscales: the Positive subscale contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness/persecution, and hostility; the Negative subscale contains seven questions to assess blunted effect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of motivation, and similar symptoms; and the General Psychopathology subscale addresses other symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS total score is the sum of all 30 items and ranges from 30 through 210. A higher score is associated with greater illness severity.
Time Frame: Baseline and 6 week
Population: mITT (modified intent-to-treat) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Number analyzed (Participants) | 145 | 152 | 142
units on a scale | -17.9 (1.72) | -17.3 (1.67) | -13.1 (1.72)
Statistical Analysis 1: Comparison: SM-13496 (Lurasidone HCl) 40mg vs Placebo; Test type: Superiority; p = 0.050, Mixed Model for Repeated Measures; LS Mean difference = -4.8, 95% CI 2-sided [-9.52 to 0.00]
Statistical Analysis 2: Comparison: SM-13496 (Lurasidone HCl) 80mg vs Placebo; Test type: Superiority; p = 0.080, Mixed Model for Repeated Measures; LS Mean difference = -4.2, 95% CI 2-sided [-8.91 to 0.50]

2. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Severity of Illness (CGI-S) Score at Week 6
Description: CGI-S is a clinician-rated assessment of the participant's current disease state on a 7-point scale, where a higher score is associated with greater severity of the disease.
  The change from baseline in CGI-S score (repeated measures) at each visit during the treatment phase is presented for the mITT population
Time Frame: Baseline and 6 weeks
Population: mITT (modified intent-to-treat) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Number analyzed (Participants) | 140 | 150 | 138
units on a scale | -0.86 (0.100) | -0.97 (0.097) | -0.79 (0.101)
Statistical Analysis 1: Comparison: SM-13496 (Lurasidone HCl) 40mg vs Placebo; Test type: Superiority; p = 0.594, Mixed Model for Repeated Measures; LS Mean difference = -0.08, 95% CI 2-sided [-0.354 to 0.203]
Statistical Analysis 2: Comparison: SM-13496 (Lurasidone HCl) 80mg vs Placebo; Test type: Superiority; p = 0.199, Mixed Model for Repeated Measures; LS Mean difference = -0.18, 95% CI 2-sided [-0.453 to 0.095]

3. Secondary Outcome: Change From Baseline in PANSS Positive Subscale Scores at Week 6
Description: The PANSS is comprised of 30 items and three subscales. The Positive subscale contains seven questions to assess delusions, conceptual disorganization, hallucinations behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS Positive subscale score is the sum of all 7 items and ranges from 7 through 49. A higher score is associated with greater illness severity.
Time Frame: Baseline and 6 weeks
Population: mITT (modified intent-to-treat) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Number analyzed (Participants) | 145 | 152 | 142
units on a scale | -5.4 (0.54) | -6.2 (0.52) | -4.2 (0.54)
Statistical Analysis 1: Comparison: SM-13496 (Lurasidone HCl) 40mg vs Placebo; Test type: Superiority; p = 0.143, Mixed Model for Repeated Measures; LS Mean difference = -1.1, 95% CI 2-sided [-2.60 to 0.38]
Statistical Analysis 2: Comparison: SM-13496 (Lurasidone HCl) 80mg vs Placebo; Test type: Superiority; p = 0.010, Mixed Model for Repeated Measures; LS Mean difference = -1.9, 95% CI 2-sided [-3.40 to -0.46]

4. Secondary Outcome: Change From Baseline in PANSS Negative Subscale Scores at Week 6
Description: The PANSS is comprised of 30 items and three subscales. The Negative subscale contains seven questions to assess blunted effect, emotional withdrawal, poor rapport, passive/apathetic social withdrawal, lack of motivation, and similar symptoms. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS Negative subscale score is the sum of all 7 items and ranges from 7 through 49. A higher score is associated with greater illness severity.
Time Frame: Baseline and 6 weeks
Population: mITT (modified intent-to-treat) population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Number analyzed (Participants) | 145 | 152 | 142
units on a scale | -3.9 (0.46) | -3.4 (0.45) | -2.9 (0.46)
Statistical Analysis 1: Comparison: SM-13496 (Lurasidone HCl) 40mg vs Placebo; Test type: Superiority; p = 0.116, Mixed Model for Repeated Measures; LS Mean difference = -1.0, 95% CI 2-sided [-2.27 to 0.25]
Statistical Analysis 2: Comparison: SM-13496 (Lurasidone HCl) 80mg vs Placebo; Test type: Superiority; p = 0.388, Mixed Model for Repeated Measures; LS Mean difference = -0.5, 95% CI 2-sided [-1.80 to 0.70]

5. Secondary Outcome: Change From Baseline in PANSS General Psychopathology Subscale Scores at Week 6
Description: The PANSS is comprised of 30 items and three subscales. The General Psychopathology subscale addresses other 16 symptoms such as anxiety, somatic concern, and disorientation. An anchored Likert scale from 1-7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. The PANSS General Psychopathology subscale score is the sum of all 16 items and ranges from 16 through 112. A higher score is associated with greater illness severity.
Time Frame: Baseline and 6 weeks
Population: mITT (modified intent-to-treat) population
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Number analyzed (Participants) | 145 | 152 | 142
units on a scale | -8.8 (0.85) | -7.9 (0.83) | -6.3 (0.85)
Statistical Analysis 1: Comparison: SM-13496 (Lurasidone HCl) 40mg vs Placebo; Test type: Superiority; p = 0.036, Mixed Model for Repeated Measures; LS Mean difference = -2.5, 95% CI 2-sided [-4.87 to -0.17]
Statistical Analysis 2: Comparison: SM-13496 (Lurasidone HCl) 80mg vs Placebo; Test type: Superiority; p = 0.174, Mixed Model for Repeated Measures; LS Mean difference = -1.6, 95% CI 2-sided [-3.93 to 0.72]

6. Secondary Outcome: Proportion of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Proportion of participants with treatment-emergent adverse events. An adverse event was defined as any untoward medical occurrence in a patient treated with a medicinal (investigational) product and which did not necessarily have a causal relationship with this treatment. Treatment-emergent adverse events (TEAEs) were defined as adverse events with a start date on or after the date of the first dose through the end of follow-up, or adverse events occurring before the date of first dose and worsening during the treatment or follow-up period.
Time Frame: From Baseline to 6 weeks
Population: Safety population defined as subjects who receive at least one dose of the study drug in the treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Number analyzed (Participants) | 150 | 154 | 151
Participants | 103 | 107 | 97

7. Secondary Outcome: Proportion of Participants With TEAEs Leading to Discontinuation
Time Frame: From Baseline to 6 weeks
Population: Safety population defined as subjects who receive at least one dose of the study drug in the treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Number analyzed (Participants) | 150 | 154 | 151
Participants | 11 | 11 | 16

8. Secondary Outcome: Proportion of Participants With Treatment-emergent Serious Adverse Events (SAEs)
Description: Proportion of participants with treatment-emergent adverse events. A serious adverse event was defined as an AE that met one or more of the following criteria: Resulted in death; Was life-threatening (i.e., a patient was at immediate risk of death at the time of the event, not an event where occurrence in a more severe form might have caused death); Required hospitalization or prolongation of existing hospitalization; Resulted in persistent or significant disability or incapacity; Was a congenital anomaly or birth defect; Was an important medical event that might jeopardize the patient or might require medical intervention to prevent one of the outcomes listed above.
Time Frame: From Baseline to 6 weeks
Population: Safety population defined as subjects who receive at least one dose of the study drug in the treatment phase.
Measure: Count of Participants; unit: Participants
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Number analyzed (Participants) | 150 | 154 | 151
Participants | 4 | 3 | 3

ADVERSE EVENTS:
Time Frame: From Baseline to 6 weeks
Description: TEAEs were defined as adverse events (AEs) with a start date on or after the date of the first dose through the end of follow-up, or AEs occurring before the date of first dose and worsening during the treatment or follow-up period. Both TEAEs and treatment-emergent serious AEs are presented for the safety population defined as subjects who receive at least one of the study drug in the treatment phase.
  Patients experiencing multiple AEs are counted once in each category.
Arm/Group | SM-13496 (Lurasidone HCl) 40mg | SM-13496 (Lurasidone HCl) 80mg | Placebo
Serious Adverse Events (participants affected / at risk) | 4/150 | 3/154 | 3/151
Other Adverse Events (participants affected / at risk) | 99/150 | 104/154 | 94/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SM-13496 (Lurasidone HCl) 40mg (N=150) | SM-13496 (Lurasidone HCl) 80mg (N=154) | Placebo (N=151)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 3 | 3 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SM-13496 (Lurasidone HCl) 40mg (N=150) | SM-13496 (Lurasidone HCl) 80mg (N=154) | Placebo (N=151)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1
Eye pain (Eye disorders) | 2 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 1 | 1
Eye discharge (Eye disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 1
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 12 | 7
Constipation (Gastrointestinal disorders) | 13 | 5 | 12
Vomiting (Gastrointestinal disorders) | 9 | 9 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 4 | 4
Toothache (Gastrointestinal disorders) | 3 | 4 | 3
Abdominal discomfort (Gastrointestinal disorders) | 1 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 3
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 3 | 1
Cheilitis (Gastrointestinal disorders) | 2 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 1
Dyskinesia oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 2
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Tooth disorder (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Anal skin tags (Gastrointestinal disorders) | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1
Functional gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 1
Periproctitis (Gastrointestinal disorders) | 0 | 0 | 1
Chest discomfort (General disorders) | 3 | 1 | 0
Irritability (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 1 | 1
Pyrexia (General disorders) | 1 | 1 | 3
Thirst (General disorders) | 1 | 1 | 1
Application site pruritus (General disorders) | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 9 | 11 | 7
Upper respiratory tract infection (Infections and infestations) | 3 | 3 | 2
Urinary tract infection (Infections and infestations) | 2 | 2 | 1
Cellulitis (Infections and infestations) | 1 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 1 | 0
Tinea infection (Infections and infestations) | 0 | 1 | 1
Tinea pedis (Infections and infestations) | 1 | 0 | 2
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Abscess (Infections and infestations) | 0 | 0 | 1
Adenoviral conjunctivitis (Infections and infestations) | 0 | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 0 | 1
Gingival infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tooth avulsion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bone fissure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Weight decreased (Investigations) | 2 | 3 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 0 | 1 | 0
Monocyte count increased (Investigations) | 1 | 0 | 0
Protein urine present (Investigations) | 0 | 1 | 0
Skin test positive (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2
Blood potassium increased (Investigations) | 0 | 0 | 1
Electrocardiogram PR shortened (Investigations) | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 2
Urobilinogen urine increased (Investigations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Polydipsia (Metabolism and nutrition disorders) | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Diet refusal (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Akathisia (Nervous system disorders) | 11 | 16 | 5
Headache (Nervous system disorders) | 14 | 6 | 12
Somnolence (Nervous system disorders) | 9 | 4 | 1
Tremor (Nervous system disorders) | 5 | 8 | 4
Dystonia (Nervous system disorders) | 4 | 6 | 1
Dizziness (Nervous system disorders) | 2 | 2 | 1
Dyskinesia (Nervous system disorders) | 1 | 3 | 1
Bradykinesia (Nervous system disorders) | 1 | 2 | 0
Extrapyramidal disorder (Nervous system disorders) | 3 | 0 | 0
Dysarthria (Nervous system disorders) | 2 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 2 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Tardive dyskinesia (Nervous system disorders) | 1 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 11 | 11 | 8
Insomnia (Psychiatric disorders) | 10 | 11 | 6
Schizophrenia (Psychiatric disorders) | 6 | 6 | 12
Psychotic disorder (Psychiatric disorders) | 3 | 1 | 4
Agitation (Psychiatric disorders) | 0 | 4 | 3
Sleep disorder (Psychiatric disorders) | 2 | 1 | 2
Aggression (Psychiatric disorders) | 2 | 0 | 0
Intentional self-injury (Psychiatric disorders) | 0 | 2 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Impulse-control disorder (Psychiatric disorders) | 1 | 0 | 0
Persecutory delusion (Psychiatric disorders) | 1 | 0 | 0
Psychiatric symptom (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1
Withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0
Catatonia (Psychiatric disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Self injurious behaviour (Psychiatric disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 1 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 4 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scar pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0
Wisdom teeth removal (Surgical and medical procedures) | 1 | 0 | 0
Hypertension (Vascular disorders) | 2 | 1 | 4
Hypotension (Vascular disorders) | 0 | 1 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes